CLINICAL TRIAL: NCT04269889
Title: Treatment of Refractory Diamond-Blackfan Anemia With Eltrombopag
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200021; 20-H-0021
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-11

CONDITIONS: Anemia, Diamond-Blackfan
Keywords: Chelation, Ribosomopathy; Erythroid Aplasia; Iron Homeostasis; Hemoglobin Synthesis; Heme Synthesis
MeSH Terms: conditions — Anemia, Diamond-Blackfan; Anemia, Aplastic | interventions — eltrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Refractory Diamond-Blackfan Anemia in Eltrombopag (Experimental): Participants with Refractory Diamond-Blackfan Anemia will be administered Eltrombopag. Participants 12 years of age an above will receive the adult dose of 150 mg by mouth daily. Participants between ages of 6 and 11 years old will start at 75 mg by mouth daily, and children 2 and 5 years of age will start at 2.5 mg/kg, not to exceed 75 mg by mouth daily.
  To adjust for the higher expected exposure in participants of East Asian and South East Asian ancestry, the starting dose for East Asian and South East Asian participants 12 years of age and above will be 75 mg by mouth once daily. For East Asian and South East Asian participants between 6 and 11 years of age, the starting dose will be 37.5 mg once daily by mouth, and for children between 2 and 5, the starting dose will be 1.25 mg/kg by mouth.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag will be administered to participants 12 years of age an above will receive the adult dose of 150 mg by mouth daily. Participants between ages of 6 and 11 years old will start at 75 mg by mouth daily, and children 2 and 5 years of age will start at 2.5 mg/kg, not to exceed 75 mg by mouth daily.
  To adjust for the higher expected exposure in participants of East Asian and South East Asian ancestry, the starting dose for East Asian and South East Asian participants 12 years of age and above will be 75 mg by mouth once daily. For East Asian and South East Asian participants between 6 and 11 years of age, the starting dose will be 37.5 mg once daily by mouth, and for children between 2 and 5, the starting dose will be 1.25 mg/kg by mouth.
  Other Names: EPAG

SUMMARY:
Background:

Diamond-Blackfan anemia (DBA) is treated with steroids. But some people cannot take steroids, or steroids don t work. Other patients must get blood transfusions regularly which are time consuming and can have significant side effects. The drug eltrombopag can increase red blood cells. Researchers want to see if it can help people with DBA and, if so, for how long.

Objective:

To study the safety and efficacy of eltrombopag in people with DBA who have not responded to steroids or could not take them.

Eligibility:

People ages 2 and older with DBA who did not respond to steroids or could not take them, or their disease has returned despite taking them

Design:

Participants will be screened with:

Medical and medicine history

Physical exam

MRI: Participants will lie in a machine that takes pictures of the liver.

Blood and urine tests

Bone marrow biopsy: A thin needle will remove a marrow sample from the participant's hip bone.

Electrocardiogram

Participants will take eltrombopag pills once daily for 24 weeks. They will have blood taken every 2 weeks.

Participants will have visits 6 months. At 6 months, they will repeat all the screening tests and also have:

Quality-of-life questionnaire

Neurodevelopmental test (for participants younger than 18 years)

If participants blood cell counts improve, they may keep taking eltrombopag for up to 3 more years. If so, they will have blood taken every 4 weeks. They will visit NIH every 6 months and repeat the above tests.

Participants will be monitored for up to 3 years after they stop taking eltrombopag. They will visit NIH 6 months after treatment ends. If participants blood counts go down after treatment ends, they may restart the drug....

DETAILED DESCRIPTION:
Diamond-Blackfan anemia (DBA) is a heritable bone marrow failure (BMF) syndrome characterized by selective erythroid defects typically presenting within the first year of life as a normochromic, macrocytic anemia with reticulocytopenia. More than half of all DBA cases are associated with either inherited or spontaneous mutations in ribosomal proteins, making DBA a prototypic ribosomopathy. Furthermore, although the primary presentation is isolated anemia, as life expectancy has improved, progressive defects in other lineages have now been identified, consistent with a long-term stem cell defect. Current standard of care for DBA is the use of systemic corticosteroids, the mechanism of which is unclear, although only half show an initial response. Even when a response to steroids is observed, long-term steroid therapy carries significant morbidity, especially in children or in combination with transfusion-associated iron overload, and thus most cannot tolerate high-dose steroids long-term. Responses are rare with second-line immunomodulatory agents. Yet other than allogeneic hematopoietic stem cell transplantation in those patients with healthy matched donors, there are no alternative therapies.

In one model for DBA pathogenesis, the defects lead to an overabundance of the iron-carrying moiety heme in primitive erythroid cells, unbound by protein. Free heme is toxic to cells, likely exacerbated over time by iron overload due to transfusions. Ongoing work with eltrombopag (EPAG) has shown that it is capable of acting as a potent iron chelator, including intracellular iron, with evidence that this effect of EPAG can reverse the impact of excess heme and elevated reactive oxygen species. Furthermore, in a recent trial of EPAG for moderate aplastic anemia or hypoproliferative unilineage cytopenias, we identified a robust response to EPAG in the one DBA patient enrolled in this clinical trial. This response has been durable over more than three years since study entry, but requires continuous EPAG to maintain transfusion independence. From these data, we hypothesize that EPAG may be able to improve production of red blood cells in DBA patients via chelation of iron and subsequent reduction in heme synthesis, resulting in decreased toxicity to bone marrow stem cells and developing erythroid cells.

We will conduct a single-arm, pilot trial in patients with steroid-refractory or steroid-intolerant DBA, treating with a fixed dose of EPAG for 6 months to assess safety and efficacy at improving hematological manifestations of DBA. Responders at 6 months will be able to continue EPAG on the extension part of this protocol for an additional 3 years. We will examine the hematologic, molecular, cytogenetic and clonal responses to EPAG in responders and non-responders alike. Translational studies will examine the mechanism of activity of EPAG in DBA through its effects on iron metabolism, erythroid differentiation, apoptosis, global transcriptome and TPO signaling pathways in patient's hematopoietic stem and progenitor cells (HSPCs).

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be participate in this study, individuals must meet all of the following criteria:

* Diamond-Blackfan anemia defined as anemia presenting on or before the third year of life with reticulocytopenia and greatly reduced or absent bone marrow erythroid precursors, supported by, but not requiring either:

  * familial history
  * gene mutation testing demonstrating a known disease-causing mutation or a mutation of disease-associated gene in combination with clinical characteristics of DBA
* Patients with late-onset DBA (diagnosed after the third year of life) may also be included if gene mutation testing confirms a disease -causing mutation as above.
* Clinically-significant anemia as defined as either:

  * hemoglobin less than 9.0 g/dL
  * red cell transfusion of at least 2 units PRBC for adults or 30 cc/kg for children (whichever is less) in the eight weeks prior to study enrollment
* Relapsed and/or steroid-refractory or intolerant of systemic corticosteroids
* Age greater than or equal to 2 years
* Weight greater than or equal to 12 kilograms
* Residence within the United States of America or territories, or able to reside within the US or its territories while on drug during trial participation

EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will not be eligible for participation in this study. However, having met exclusion criteria in the past does not preclude study participation if the criteria are no longer met, unless otherwise specified (i.e. patients with modifiable factors such as laboratory abnormalities or acute health problems may be re-screened). For laboratory assessments, this requires no less than two weeks from the previous exclusionary finding. The intervals for health problems that must elapse prior to re-screening are specified below.

* Platelet count > 400,000 / microliter
* Stage 4 or greater kidney disease as defined by creatinine > 2.5 mg/ dL or GFR < 30 mL/min/1.73 m(2)

  --For pediatric patients 17-years-old or younger, GFR shall be used. This can be estimated using the bedside Schwartz equation, the Counahan-Barratt method, or a similar methodology. Direct measurement including, but not limited to, 24-hour urine creatinine clearance or radiographic methods is recommended for patients with stage 3 disease (GFR less than or equal to 45 mL/min/1.73 m(2)).
* Direct bilirubin > 2.0 mg/ dL, including congenital abnormalities in the bilirubin level
* SGOT (AST) or SGPT (ALT) > 5 times the upper limit of normal
* Treatment with androgens (danazol or oxymetholone) or corticosteroids less than 4 weeks prior to initiating eltrombopag.

  --Physiologic steroid replacement for adrenal insufficiency or other similar conditions is not exclusive of trial participation
* Treatment with any medications that may interfere with the metabolism of eltrombopag (e.g., CYP1A2 and CYP2C8 modulators) or whose own altered metabolism by eltrombopag cannot be adjusted for
* Hypersensitivity to eltrombopag or its components
* Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient s ability to tolerate protocol therapy, or that death within 7-10 days is likely
* Life expectancy of less than 3 months for any cause
* Subjects with known liver cirrhosis in severity that would preclude tolerability of eltrombopag as evidenced by albumin < 3.5g/dL
* History or current diagnosis of cardiac disease indicating significant risk of safety for patients participating in the study such as uncontrolled or significant cardiac disease, including any of the following:

  * Recent myocardial infarction (within last 6 months),
  * Uncontrolled congestive heart failure,
  * Unstable angina (within last 6 months),
  * Clinically significant (symptomatic) cardiac arrhythmias (e.g., sustained ventricular tachycardia, and clinically significant second or third-degree AV block without a pacemaker.)
  * Long QT syndrome, family history of idiopathic sudden death, congenital long QT syndrome or additional risk factors for cardiac repolarization abnormality, as determined by the investigator
  * Impaired cardiac function such as corrected QTc>450msec using Fridericia correction on the screening EKG, other clinically significant cardio-vascular disease (e.g. uncontrolled hypertension, history of labile hypertension), history of known structural abnormalities (e.g. cardiomyopathy).
* Known active or uncontrolled infections not adequately responding to appropriate therapy.

  --HIV infection is not exclusive of trial participation if the infection is effectively controlled with medications not known to interfere with eltrombopag metabolism or be metabolized by pathways known to be altered by eltrombopag. HIV RNA viral load must be undetectable at the time of enrollment, and CD4 cell count must be greater than or equal to 200/microliter. Patients must remain on antiretroviral therapy throughout study participation and must be periodically monitored for suppression of viral load and CD4 cell count. If drug-drug interactions between antiretroviral medications and eltrombopag are suspected, these must be addressed by a qualified clinical pharmacist or pharmacologist, and any changes to antiretroviral therapy need to be approved in consultation with an Infectious Disease and/or HIV specialist prior to enrollment.
* Active malignancy or likelihood of recurrence of malignancies within 12 months
* Evidence for MDS or AML as defined by WHO criteria.
* Patients who have received chemotherapeutic treatment or other specific antineoplastic drugs or radiation therapy within 6 months of study entry
* Female subjects who are nursing or pregnant (positive serum or urine beta-human chorionic gonadotrophin (b-hCG) pregnancy test) at screening or pre-dose on Day 1.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 30 days after the last dose of eltrombopag. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to screening). For female patients on the study the vasectomized male partner should be the sole partner for that patient.
  * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
  * In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
  * Women are considered post-menopausal and not of child bearing potential if they have had over 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile age appropriate (e.g. generally 40-59 years), history of vasomotor symptoms (e.g. hot flushes) in the absence of other medical justification or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment should she be considered not of child bearing potential.

    * Sexually active males unless they use a condom during intercourse while taking the study treatment and for 30 days after stopping study treatment and should not father a child in this period. A condom is required to be used also by vasectomized men as well as during intercourse with a male partner in order to prevent delivery of the drug via seminal fluid.
* History of thromboembolic events other than catheter-related thromboses
* Active alcohol/drug abuse
* Unable to understand the investigational nature of the study or give informed consent and does not have a legally authorized representative or surrogate that can provide informed consent
* Unable to take investigational drug
* Concurrent participation in an investigational study within 30 days prior to enrollment or within 5-half-lives of the investigational product, whichever is longer. Note: parallel enrollment in a disease registry is permitted.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2024-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Young, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-H-0021.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled from February 2020 through August 2022 at the National Institutes of Health (NIH) (Bethesda, MD).
Period: Initial Phase (Day 0 to Month 6)
Arm/Group | Refractory Diamond-Blackfan Anemia in Eltrombopag
Started | 15
Completed | 1
Not Completed | 14
Not completed — Lack of Efficacy | 14
Period: Extended Phase (6 Months to Year 3)
Arm/Group | Refractory Diamond-Blackfan Anemia in Eltrombopag
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Refractory Diamond-Blackfan Anemia in Eltrombopag
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Number of participants with Iron Overload [Count of Participants; unit: Participants] | 14

OUTCOME MEASURES:

1. Primary Outcome: Participants That Responded to Eltrombopag
Description: Participants that responded to Eltrombopag as defined by:
  Response to treatment will be defined by one or more of the following:
  * Erythroid response for subjects with a pretreatment hemoglobin less than 9 G/dL will be defined as an increase in hemoglobin by >1.5 G/dL from enrollment baseline, and/or
  * A reduction in the units of PRBC transfusions by at least 50% during the eight consecutive weeks prior to response assessment - compared with the pretreatment transfusion number in the previous 8 weeks.
Time Frame: 6 months (24 weeks +/- 14 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Refractory Diamond-Blackfan Anemia in Eltrombopag
Number analyzed (Participants) | 15
Participants
  Response to Treatment | 1
  No Response to Treatment | 14

2. Primary Outcome: Time (Weeks) to Response
Description: Time-to-response in weeks will also be measured according to the time from Eltrombopag initiation to the first time the patient met criteria for response.
  Response to treatment will be defined by one or more of the following:
  * Erythroid response for subjects with a pretreatment hemoglobin less than 9 G/dL will be defined as an increase in hemoglobin by >1.5 G/dL from enrollment baseline, and/or
  * a reduction in the units of PRBC transfusions by at least 50% during the eight consecutive weeks prior to response assessment - compared with the pretreatment transfusion number in the previous 8 weeks.
Time Frame: 6 months (24 weeks +/- 14 days)
Population: Analysis includes only participants that responded to eltrombopag
Measure: Number; unit: weeks
Arm/Group | Refractory Diamond-Blackfan Anemia in Eltrombopag
Number analyzed (Participants) | 1
weeks | 15

3. Primary Outcome: Number of Adverse Events
Description: Number of Adverse Events
  Toxicity profile as measured by using the Common Terminology Criteria for Adverse Events (CTCAE version 5.0) for grade 2 and above. According to https://ctep.cancer.gov/, CTCAE is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. CTCAE grades are defined as:
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental activities of daily living.
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4 Life-threatening consequences; urgent intervention indicated.
Time Frame: 6 months (24 weeks +/- 14 days)
Population: Analysis includes number of adverse events with grade 2 events and above
Measure: Number; unit: Adverse Events
Groups:
- Refractory Diamond-Blackfan Anemia in Eltrombopag With Grade 2 Adverse Events; Refractory Diamond-Blackfan Anemia in Eltrombopag With Grade 3 Adverse Events; Refractory Diamond-Blackfan Anemia in Eltrombopag With Grade 4 Adverse Events: Participants with Refractory Diamond-Blackfan Anemia will be administered Eltrombopag. Participants 12 years of age an above will receive the adult dose of 150 mg by mouth daily. Participants between ages of 6 and 11 years old will start at 75 mg by mouth daily, and children 2 and 5 years of age will start at 2.5 mg/kg, not to exceed 75 mg by mouth daily.
  To adjust for the higher expected exposure in participants of East Asian and South East Asian ancestry, the starting dose for East Asian and South East Asian participants 12 years of age and above will be 75 mg by mouth once daily. For East Asian and South East Asian participants between 6 and 11 years of age, the starting dose will be 37.5 mg once daily by mouth, and for children between 2 and 5, the starting dose will be 1.25 mg/kg by mouth.
Arm/Group | Refractory Diamond-Blackfan Anemia in Eltrombopag With Grade 2 Adverse Events | Refractory Diamond-Blackfan Anemia in Eltrombopag With Grade 3 Adverse Events | Refractory Diamond-Blackfan Anemia in Eltrombopag With Grade 4 Adverse Events
Number analyzed (Participants) | 15 | 15 | 15
Adverse Events
  Headache | 0 | 2 | 0
  Arthralgia | 1 | 1 | 0
  Back pain | 1 | 0 | 0
  Chills | 1 | 1 | 0
  Dysphagia | 1 | 0 | 0
  Fever | 1 | 1 | 0
  Flu-like symptoms: COVID/flu | 0 | 1 | 0
  Elevated alanine transaminase | 0 | 1 | 0
  Acute inception without sepsis/Acute viral syndrome | 1 | 0 | 0
  Myalgia | 1 | 0 | 0
  Nausea | 0 | 1 | 0
  Sepsis | 0 | 1 | 0

4. Secondary Outcome: Number of Participants That Responded to Eltrombopag
Description: Number of Participants That Responded to Eltrombopag. As determined by the response to treatment, which will be assessed based on one or more of the following criteria:
  Erythroid response for subjects with a pretreatment hemoglobin less than 9 G/dL will be defined as an increase in hemoglobin by >1.5 G/dL from enrollment baseline, and/or
  A reduction in the units of PRBC transfusions by at least 50% during the eight consecutive weeks prior to response assessment - compared with the pretreatment transfusion number in the previous 8 weeks.
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Refractory Diamond-Blackfan Anemia in Eltrombopag
Number analyzed (Participants) | 15
Participants
  Response to Treatment | 0
  No Response to Treatment | 15

5. Secondary Outcome: Number of Participants With Robust Response to Eltrombopag
Description: Number of Participants with Robust Response to Eltrombopag regardless when it is achieved. Best response is defined as robust response or not robust response.
  Robust response to treatment will be defined both:
  * Stable hemoglobin (two consecutive measurements at least 2 weeks apart) greater than 10 g/dL, and
  * Transfusion independence for the previous 8 weeks
Time Frame: 3 Months, 6 Months, Up to 27 Months
Population: Analysis post 6 months only includes those participants that met criteria for extension phase of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Refractory Diamond-Blackfan Anemia in Eltrombopag
Number analyzed (Participants) | 15
Participants
  3 months : Robust Response | 0
  3 months : Not Robust Response | 15
  6 months : Robust Response | 0
  6 months : Not Robust Response | 15
  Up to 27 months : Robust Response: number analyzed (Participants) | 1
  Up to 27 months : Robust Response | 0

6. Secondary Outcome: Median Change in Platelet Count
Description: Median Change in Platelet Count as measured by serial CBC assessments
Time Frame: Baseline, 3 months
Population: Analysis includes those participants that completed baseline and month 3 visits
Measure: Median (Full Range); unit: K/uL
Arm/Group | Refractory Diamond-Blackfan Anemia in Eltrombopag
Number analyzed (Participants) | 12
K/uL | 83.0 [-10.0 to 432.0]

7. Secondary Outcome: Median Change Absolute Neutrophil Count
Description: Median Change Absolute Neutrophil Count as measured by serial CBC assessments
Time Frame: Baseline, Month 3
Population: Analysis includes those participants that completed baseline and month 3 visits
Measure: Median (Full Range); unit: K/uL
Arm/Group | Refractory Diamond-Blackfan Anemia in Eltrombopag
Number analyzed (Participants) | 12
K/uL | 0.7 [-2.6 to 4.2]

8. Secondary Outcome: Number of Participants That Experienced Relapse
Description: Number of Participants that experienced Relapse during extension phase. Relapse is defined as no longer meeting response criteria.
  Response criteria is defined as: Response to treatment will be defined by one or more of the following:
  * Erythroid response for subjects with a pretreatment hemoglobin less than 9 G/dL will be defined as an increase in hemoglobin by >1.5 G/dL from enrollment baseline, and/or
  * A reduction in the units of PRBC transfusions by at least 50% during the eight consecutive weeks prior to response assessment - compared with the pretreatment transfusion number in the previous 8 weeks.
Time Frame: 6 months up to 27 months
Population: All participants that participated within the extended phase of the clinical trial
Measure: Count of Participants; unit: Participants
Arm/Group | Refractory Diamond-Blackfan Anemia in Eltrombopag
Number analyzed (Participants) | 1
Participants | 0

9. Secondary Outcome: Number of Participants That Experienced Clonal Evolution
Description: Number of participants that experienced clonal evolution according to cytogenetic, mutational or flow cytometric markers
Time Frame: 6 Months and Up to 27 months
Population: Analysis post 6 months only includes those participants that met criteria for extension phase of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Refractory Diamond-Blackfan Anemia in Eltrombopag
Number analyzed (Participants) | 15
Participants
  6 months | 0
  Up to 27 months: number analyzed (Participants) | 1
  Up to 27 months | 1

10. Secondary Outcome: Number of Adverse Events During the Extension Phase
Description: as for outcome 3
Time Frame: 6 months Up to 27 months
Population: All participants that participated within the extended phase of the clinical trial
Measure: Number; unit: Adverse Events
Arm/Group | Refractory Diamond-Blackfan Anemia in Eltrombopag
Number analyzed (Participants) | 1
Adverse Events
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0
  Grade 5 | 0

11. Secondary Outcome: Neurodevelopment in Pediatric Patients
Description: Neurodevelopment in pediatric patients as measured by validated neurodevelopmental measurements
Time Frame: At baseline and Month 6
Population: Data was not collected and there are no future plans to collect the data. The analysis could not be completed due to insufficient staffing to carry out the required tasks.
Arm/Group | Refractory Diamond-Blackfan Anemia in Eltrombopag
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants With Iron Overload
Description: Number of participants with Iron overload. Iron overload as measured by serial ferritin levels, T2* MRI measurements and bone marrow iron staining
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Refractory Diamond-Blackfan Anemia in Eltrombopag
Number analyzed (Participants) | 15
Participants | 15

ADVERSE EVENTS:
Time Frame: up to 27 months
Description: Grade 2 adverse events and above, including clinically significant abnormal non-hematologic findings on laboratory evaluations, regardless of severity and attribution, will be recorded at each study visit and followed until satisfactory resolution.
Arm/Group | Refractory Diamond-Blackfan Anemia in Eltrombopag
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 2/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Refractory Diamond-Blackfan Anemia in Eltrombopag (N=15)
Nausea (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Elevated alanine transaminase (Hepatobiliary disorders) | 1 (1)
Flu like symptoms (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Refractory Diamond-Blackfan Anemia in Eltrombopag (N=15)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Acute inception without sepsis/Acute viral syndrome (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT04269889/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT04269889/ICF_000.pdf